CLINICAL TRIAL: NCT02544139
Title: Determination of Estimated Specificity of Chagas Detect Plus Rapid Tests
Brief Title: Specificity Study of Diagnostic for Chagas Disease
Status: Completed | Type: Observational
Sponsor: InBios International, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DSC0227
Record Dates: First submitted 2015-09-04; First posted 2015-09-09 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Infectious Diseases
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum

INTERVENTIONS:
Other: Chagas Detect Plus

SUMMARY:
This study assesses the specificity of Chagas Detect™ Plus (CDP) rapid test versus standard reference tests (e.g. RIPA or IFA) for Chagas diagnosis in the US.

The Chagas Detect™ Plus Rapid Test is a rapid immunochromotagraphic strip assay for the qualitative detection of antibodies to Trypanosoma cruzi (T. cruzi) in human serum or whole blood samples. Reactive assay results are presumptive evidence of Chagas infection.

This study will enroll males and females 18-70 years of age from areas non-endemic for Chagas infection. A fingerprick blood sample and a venous blood sample (for processing to serum) will be collected from each subject. Subject age, gender, and symptoms will be recorded. For this study, samples will have no personally identifiable information.

CDP and reference tests will be performed by different operators who are laboratory staff members. These staff members, blinded to each other's results, will evaluate the samples from each method independently.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects 18 to 70 years of age
2. Subjects must be able to answer questions concerning:

   1. Clinical symptoms
   2. Blood transfusions
   3. Organ transplants
   4. Travel or residence in Chagas endemic areas

Exclusion Criteria:

1. Any subject who knows that they have positive serology for Chagas disease
2. Subjects who are unable to understand verbal of written or oral language of the consent, or require a legal authorized representative for consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will enroll male and female subjects between 18 and 70 years of age without known risk factors for Chagas. Typically Chagas disease is a chronic, asymptomatic disease.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
number of subjects with negative result | one day

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States